CLINICAL TRIAL: NCT00005495
Title: Primary Prevention of CHD Risk Factors Occurring in US
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5013; R03HL058697 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Heart Disease Risk Reduction; Coronary Disease; Hypertension; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension; Hypercholesterolemia

SUMMARY:
To evaluate the effectiveness of primary prevention of coronary heart disease risk factors by examining data from the National Health Examination Survey (NHES) and the National Health and Nutrition Examination Surveys (NHANES) to determine whether more recent birth cohorts were attaining lower blood pressure and cholesterol levels than earlier birth cohorts.

DETAILED DESCRIPTION:
BACKGROUND:

The coronary heart disease risk factor profile of Americans has been improving, with decreasing blood pressure and cholesterol levels. However, it is not apparent whether this improvement is due to primary prevention of risk factors through lifestyle choices or to secondary prevention (management) of established risk factors. Since secondary prevention only targets people with high blood pressure or cholesterol levels, the effect should be demonstrated by temporal declines in the upper percentiles (75th, 90th) of the blood pressure and cholesterol distributions. Primary prevention should shift the entire risk factor distribution, including the percentiles in the middle (50th) and lower (10th, 25th) portions of the distribution. Thus, the effectiveness of primary prevention programs can be evaluated by examining temporal changes in the middle and lower percentiles, and the effectiveness of secondary prevention can be evaluated by examining temporal changes in the higher percentiles.

DESIGN NARRATIVE:

Data from the National Health Examination Survey and the National Health and Nutrition Examination Surveys were examined to determine whether more recent birth cohorts were attaining lower blood pressure and cholesterol levels than earlier birth cohorts. The results of these analyses provided information that may help guide further research and application of population prevention strategies.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-07; Study Completion 1999-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Goff, Jr. — Wake Forest University

REFERENCES:
- [Background] Goff DC Jr, Labarthe DR, Howard G, Russell GB. Primary prevention of high blood cholesterol concentrations in the United States. Arch Intern Med. 2002 Apr 22;162(8):913-9. doi: 10.1001/archinte.162.8.913. PMID 11966343
- [Background] Goff DC, Howard G, Russell GB, Labarthe DR. Birth cohort evidence of population influences on blood pressure in the United States, 1887-1994. Ann Epidemiol. 2001 May;11(4):271-9. doi: 10.1016/s1047-2797(00)00224-6. PMID 11306346